CLINICAL TRIAL: NCT00569257
Title: Antitumoral Activity and Safety of AEZS-108 (AN-152), a LHRH Agonist Linked Doxorubicin, in Women With LHRH Receptor Positive Gynecological Tumors
Brief Title: Antitumoral Activity and Safety of AEZS-108 in Women With LHRH Receptor Positive Gynecological Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AEterna Zentaris (Industry)
Collaborators: AGO Study Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AEZS-108-040; AGO-GYN 5; EudraCT No. 2007-002663-26
Record Dates: First submitted 2007-12-06; First posted 2007-12-07 (Estimated); Last update posted 2011-12-13 (Estimated); Status verified 2011-12

CONDITIONS: Ovarian Cancer; Endometrial Cancer
Keywords: LHRH receptor; receptor positive tumors; platinum resistant ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms | interventions — LHRH, lysine(6)-doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: AEZS-108 — intravenous infusion at a dose of 267 mg/sqm every 3 weeks, up to 6 treatment cycles
  Other Names: AN-152

SUMMARY:
The purpose of this study is to determine whether AEZS-108 shows anti-tumor activity and is tolerated in patients with gynecological tumors (ovarian / endometrial cancer) that have been shown to express receptors for the luteinizing hormone releasing hormone (LHRH)

DETAILED DESCRIPTION:
The ovary and the endometrium are hormone dependent organs. Receptors for different sex hormones are found commonly in epithelial ovarian and endometrial cancers. LHRH and its receptors are expressed in about 80% of human ovarian and endometrial cancers. As binding sites are present on tumors in higher concentrations than on most normal tissues, these receptors represent a specific target for AEZS-108 in which doxorubicin is coupled to an LHRH analog.

Patients whose tumor specimen have shown to be positive for LHRH receptor expression will be investigated for tumor response and tolerability.

ELIGIBILITY:
Inclusion Criteria:

* LHRH receptor positive tumor status: positive receptor status determined by immunohistochemistry from primary tumor
* Histologically confirmed epithelial ovarian cancer (Stratum A)
* Advanced (FIGO III or IV) or recurrent disease
* Progression during treatment with a platinum-based regimen or within 6 months after receiving a platinum-based regimen
* Previous treatment with a taxane-containing regimen
* At least one measurable target lesion (RECIST criteria) OR CA125 level higher than twice the upper limit of normal range (GCIG criteria)
* Histologically confirmed endometrial cancer (Stratum B)
* Advanced (FIGO III or IV) or recurrent disease not amenable to potentially curative treatment with local surgery and/or radiation therapy
* No previous anthracycline-based chemotherapy
* At least one measurable target lesion according to RECIST criteria

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2007-12; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Tumor response as per RECIST or (for Ovarian CA patients without evaluable target lesion following RECIST) GCIG criteria | up to six 3-weekly treatment cycles

SECONDARY OUTCOMES:
Time-to-progression (TTP); Overall survival | up to observation of event
Safety of AEZS-108 (possibly drug-related adverse events) | 4 weeks beyond last drug admnistration

CONTACTS AND LOCATIONS:
Overall Officials: Günter Emons, Prof.Dr.med., Principal Investigator — Universitäts-Frauenklinik / Department of Obstetrics and Gynecology, University of Göttingen
Locations (17):
- Bulgaria (3):
  - University Hospital "Dr. Georgy Stranski", Pleven
  - Regional Oncology Hospital Plovdiv, Plovdiv
  - Regional Oncodispensary "M.Markov", Varna
- Germany (14):
  - Klinik für Frauenheilkunde und Geburtshilfe, Charité Campus Virchow-Klinikum, Berlin
  - Frauenklinik, Klinikum Bremen-Mitte GmbH, Bremen
  - Klinik für Frauenheilkunde und Geburtshilfe, Universitätsklinikum Carl Gustav Carus, Dresden
  - Klinik für Frauenheilkunde, Universität Erlangen-Nürnberg, Erlangen
  - Universitätsfrauenklinik, Universitätsklinikum, Essen
  - Universitätsfrauenklinik, Klinikum der JWG Universität Frankfurt, Frankfurt am Main
  - Frauenklinik, Georg-August-Universität Göttingen, Göttingen
  - Klinikum der Ernst-Moritz-Arndt-Universitaet, Klinik und Poliklinik fuer Gynaekologie und Geburtshilfe, Greifswald
  - Frauenklinik, Medizinische Hochschule Hannover, Hanover
  - Frauenklinik, St. Vincentius Kliniken AG, Karlsruhe
  - Klinik für Gynäkologie und Geburtshilfe, Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Frauenklinik, Klinikum Lüneburg, Lüneburg
  - Klinikum Suedstadt der Hansestadt Rostock, Universitaetsfrauenklinik und Poliklinik, Rostock
  - Klinik f. Gynäkologie u. Gyn. Onkologie, Dr. Horst Schmidt Kliniken GmbH, Wiesbaden

REFERENCES:
- See also: AGO Studiengruppe Ovarialkarzinom — http://www.ago-ovar.de